CLINICAL TRIAL: NCT03931070
Title: The Effect of Ramelteon on Delirium and Sleep in Patients Admitted to the ICU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1364075
Record Dates: First submitted 2019-02-22; First posted 2019-04-30 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2021-09

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mechanically ventilated (Experimental): Participants who are on mechanical ventilator at the time of study enrollment.
  Interventions: Drug: Ramelteon; Drug: Placebo - Cap
- Non mechanically ventilated (Experimental): Participants who are not on mechanical ventilator at the time of study enrollment.
  Interventions: Drug: Ramelteon; Drug: Placebo - Cap

INTERVENTIONS:
Drug: Ramelteon — Patients assigned to Ramelteon group will receive 8mg of Ramelteon every night throughout the hospitalization or up to 30 days, whichever is sooner.
  Other Names: Rozerem
Drug: Placebo - Cap — Patients assigned to Placebo group will receive placebo pill that is indistinguishable from Ramelteon, every night throughout the hospitalization or up to 30 days, whichever is sooner.
  Other Names: Placebo

SUMMARY:
Delirium is a disturbance in attention and awareness that occurs over a short period of time. Delirium is common in critically ill patients, and poor sleep quality in the intensive care unit (ICU) often worsens delirium. We aim to lower delirium in the intensive care unit (ICU) by using ramelteon, which is a drug used to improve sleep at night.

DETAILED DESCRIPTION:
Rationale:

Many pharmacologic agents have been studied to reduce delirium in high risk patients, but the data has not shown significant or clinically important outcomes. These agents also have more side effect profiles such as arrhythmia and QT prolongation. Ramelteon is an effective drug to improve sleep quality and has a low side effect profile. Improved sleep quality and reduced delirium in ICU population will lead to improved acute and long-term outcomes of the patients and lower delirium-related healthcare cost.

Study Hypothesis:

It is hypothesized that those receiving ramelteon will have a higher rate of delirium- and coma-free days, on average, than those receiving placebo. We also hypothesize that those receiving ramelteon will have lower Confusion Assessment Method for Intensive Care Unit-7 (CAM-ICU-7) scores than those receiving placebo, and that the reduction from baseline will be greater for those receiving ramelteon than those receiving placebo. In addition, those receiving ramelteon will be in the medical intensive care unit (MICU) and hospital fewer days than those receiving placebo. Those receiving ramelteon will have more sleep-time and fewer awakenings than those receiving placebo (as defined by the actigraph device). In addition, those receiving ramelteon will have higher subjective quality of sleep than those receiving placebo on patient-reported sleep evaluation questionnaire. Lastly, those receiving ramelteon will suffer less from post-intensive care syndrome compared to those receiving placebo.

Study Procedure:

Every day, investigator(s) will identify patients who meet criteria on chart review and these patients will be approached for consent. Consent will be obtained by patient or surrogate decision maker as appropriate.

After consent is obtained, investigator will call pharmacy investigational service to provide patient information/patient study identification for randomization and medication allotment. Pharmacy investigational services will be informed whether the patient is mechanically ventilated or not (this is a subgroup that will require randomization in the urn randomization design). Patient's data will be recorded on REDcap including patient identification and delirium assessment. A sign will be placed at the door of the patient's room to identify patient as a study subject and to notify that the study subject should not be given ramelteon, melatonin, or fluvoxamine by the primary medical team.

Upon enrollment, patients in Ramelteon group will receive 8 mg of Ramelteon capsule nightly at 9 pm and placebo group will receive the placebo capsule. Ramelteon and Placebo capsules will be indistinguishable from each other, even when opened to be administered via nasogastric or orogastric tubes. Medication administration will continue throughout the hospital stay, with maximum of 30 days, every night until death or discharge from the hospital. If a patient's code status changes to comfort measures only, study drug administration will be discontinued.

An actigraph unit will be placed on patient's wrist for continuous non-invasive measurement of rest and activity to estimate sleep measures. The actigraph unit will be removed from the patient when the patient is discharged from the ICU. The data from the actigraph will then be extracted and analyzed by Action W software.

Patients will be assessed by investigator daily for delirium using the Confusion Method Assessment for the ICU-7 (CAM-ICU-7). For patients who are on mechanical ventilation or on sedatives, all sedative medications will be held if the primary medical team approves. CAM-ICU-7 will be performed for each patient at the time of maximal awakening and after sedation (continuous infusion and as needed doses) is held for at least 30 to 60 minutes. For those patients that are able to participate, they will complete Richmond-Campbell Sleep Questionnaire (RCSQ), which is a two minute questionnaire, to assess their previous night's sleep. The CAM-ICU-7 and RCSQ assessments will continue throughout the hospitalization after ICU discharge, until discharge from the hospital or up to 30 days. Patients will not be monitored upon discharge from the hospital (ie. discharged to nursing home, skilled nursing facility, home).

Patients will be contacted via telephone to conduct two surveys to assess post-intensive care quality of life at 1-, 3-, and 6-months after ICU discharge. Telephone Interview for Cognitive Status (TICS) will be used to assess for cognitive impairment, and EuroQol-5Dimensions (EQ-5D) will be used to assess for health quality including mobility, self-care, activity level, pain/discomfort, and anxiety/depression.

Data Safety Monitoring Plan:

We will have two faculty members from the Division of Pulmonary, Critical Care and Sleep Medicine at the Warren Alpert Medical School of Brown University as data safety monitoring members for this study in the event a study-related adverse event occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age newly admitted to ICU and expected to stay in ICU for at least three days as determined by study personnel.
* Able to take medicine via enteral access.

Exclusion Criteria:

* Taking ramelteon or fluvoxamine
* Expected life expectancy of less than 48 hours.
* Pre-existing dementia
* Alcohol withdrawal admission diagnosis
* Acute neurological condition (brain abscess/tumor, head bleed, stroke, seizure)
* Known allergy/intolerance to ramelteon
* Severe liver dysfunction: Hepatic encephalopathy, cirrhosis (Child-Pugh class C or greater)
* Suicide attempt, admission for acute psychiatric illness
* GI bleed or other inability to use enteral nutrition
* Pregnant patient
* Incarcerated
* Prior enrollment into the study
* On paralytics at the time of admission
* Unable to get enteral feeds/meds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Delirium- and coma-free days | Until discharge or up to 30 days of hospitalization, whichever is sooner.
  The average number of delirium- and coma-free days as defined by Richmond Agitation-Sedation Scale (RASS) greater than -4 (RASS score is a range from -5 to +4, the lower score indicates comatose state, the higher score indicates more awakeness/agitation) and Confusion Assessment Method in the Intensive Care Unit (CAM-ICU-7) score greater than 3 (CAM-ICU-7 score ranges from 0 to 7, the higher score indicates more severe delirium).

SECONDARY OUTCOMES:
Delirium assessment score Confusion Assessment Method-Intensive Care Unit-7 (CAM-ICU-7) in Ramelteon group compared to the placebo group. | Until discharge or up to 30 days of hospitalization, whichever is sooner.
  Confusion Assessment Method in the Intensive Care Unit (CAM-ICU-7) score will be measured to assess delirium. Score ranges from minimum 0 to maximum 7, which is obtained as a sum of each category of CAM-ICU-7 assessment, where scores 0-2 indicate no delirium and greater than 3 indicate delirium, and the higher score (greater than 3) indicates more severe delirium. Higher CAM-ICU-7 score indicates a worse outcome.
Change in the delirium assessment scores (CAM-ICU-7) from baseline score on day one of enrolment in ramelteon group compared to the placebo group. | Until discharge or up to 30 days of hospitalization, whichever is sooner.
  Confusion Assessment Method in the Intensive Care Unit (CAM-ICU-7) score will be measured to assess delirium. Score ranges from minimum 0 to maximum 7, which is obtained as a sum of each category of CAM-ICU-7 assessment, where scores 0-2 indicate no delirium and greater than 3 indicate delirium, and the higher score (greater than 3) indicates more severe delirium. Higher CAM-ICU-7 score indicates a worse outcome. Each participant's individual CAM-ICU-7 scores will be compared throughout their hospital stay to assess the presence/absence of delirium as well as its severity if delirium is present.
Number of ICU and hospital days. | Until discharge or up to 30 days of hospitalization, whichever is sooner.
  The average length of stay in the ICU and hospital, in days.
Hours of total sleep, nighttime sleep and number of awakenings in ramelteon group compared to the placebo group. | During the entire ICU stay upon enrollment up to 30 days.
  The average number of hours of sleep, and the number of awakenings as measured by actigraphy, which is a wearable accelerometer that is validated to assess sleep quality. This will be recorded during the ICU stay starting from the time of enrollment until discharge from the ICU, up to 30 days maximum.
Richards-Campbell Sleep Questionnaire (RCSQ) scores in ramelteon group compared to the placebo group. | Until discharge or up to 30 days of hospitalization, whichever is sooner.
  Richards-Campbell Sleep Questionnaire is a validated sleep survey using visual analog scale (VAS) filled out by the subject, which comprises of 5 questions with scores ranging from minimum 0 to maximum 100, which is computed as an average of the 5 subscales. The higher score indicates worse sleep quality.
Telephone Interview for Cognitive Status (TICS) scores at 1-, 3-, and 6-month post ICU discharge in ramelteon group compared to the placebo group. | At one, three, and six month post ICU discharge.
  Telephone Interview for Cognitive Status is a validated phone-based assessment of cognitive status. The score ranges from 0 to 40, which is computed as a sum of subscales. The lower score indicates worse degree of cognitive impairment.
EQ-5D (Euro Quality of life-5 Dimensions) scores at 1-, 3-, and 6-month post ICU discharge in ramelteon group compared to the placebo group. | At one, three, and six month post ICU discharge.
  Euro Quality of life-5 Dimensions is a health related quality of life questionnaire that is telephone-based. It is comprised of 5 health related quality of life questions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), and each question is in multiple-choice format. The score ranges from 5 to 25, which is computed as a sum of each subscale. The higher scores indicating worse health-related quality of life assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell M Levy, MD, MCCM, FCCP, Principal Investigator — Brown University
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No